CLINICAL TRIAL: NCT03941925
Title: Double-blind, Randomized Placebo-controlled Trial Investigating the Effect of Prebiotic Fructans on Bowel Habits of Constipated Young Children One to Three Years of Age
Brief Title: Prebiotic Fructans Effect on 1-3 Years Constipated Children's Bowel Habits
Acronym: CONSTICHILD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Beneo GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-18-016
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Constipation
Keywords: prebiotic
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic fructans (Experimental): Prebiotic fructans. Prebiotic will be mixed into foods or drinks and consumed twice daily.
  Interventions: Dietary Supplement: Prebiotic fructans
- Maltodextrin (Placebo Comparator): Maltodextrin. Maltodextrin will be mixed into foods or drinks and consumed twice daily.
  Interventions: Dietary Supplement: Non-prebiotic maltodextrin

INTERVENTIONS:
Dietary Supplement: Prebiotic fructans — Prebiotic group receiving the prebiotic fructans in two doses during the 4-week intervention period.
  Arms: Prebiotic fructans
Dietary Supplement: Non-prebiotic maltodextrin — Placebo group receiving the non-prebiotic maltodextrin in two doses during the 4-week intervention period.
  Arms: Maltodextrin

SUMMARY:
The aim of the study is to confirm the effectiveness of chicory-derived prebiotic inulin-type fructans on bowel function in young children.

DETAILED DESCRIPTION:
The aim of the study is to confirm the effectiveness of chicory-derived prebiotic inulin-type fructans on bowel function in young children. It is a double-blind, randomized, placebo-controlled trial.This study plans to recruit into the group of 100 participants (at least 80 of them completed) in 2018-2020.The two groups for the study are product group (prebiotic fructans) and control group (placebo maltodextrin).Duration of intervention is 6 weeks, including 2 weeks for run-in and 4 weeks for intervention.Efficacy parameters are stool consistency (assessed with Amsterdam infant stool scale),stool frequency, stool amount and stool color (assessed with Amsterdam infant stool scale, treatment success, tolerance and acceptability).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of functional constipation following ROME4 criteria.
2. Subject is otherwise healthy at the time of pre-examination.
3. Subject is aged 1-3 years at the time of pre-examination.
4. Subject and caretaker are able and willing to follow the study instructions.
5. Subject is suitable for participation in the study according to the investigator/physician/study personnel.
6. Written informed consent is given by parent or legal guardian.

Exclusion Criteria:

1. No legal guardian's command of any local language.
2. Organic causes of defecation disorders incl. Hirschsprung disease, Spina bifida, hypothyroidism etc.
3. Other metabolic or renal abnormalities or mental retardation (Child's mental delay).
4. Food allergies or intolerances.
5. Using drugs (e.g. antibiotics) influencing gastrointestinal function (4 weeks before run-in, 6 weeks before intervention).
6. Use of laxatives and labelled pre- and probiotics in the previous 2 weeks before the beginning of run-in (4 weeks before intervention)
7. Subjects who are currently involved or will be involved in another clinical or food study

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Stool consistency | 4 weeks
  Assessed by the parents in a continuous daily bowel diary over the study period using the Amsterdam Infant Stool Scale (AISS) comprised of a 4-point scale (A: watery, B: soft, C: formed, D: hard)

SECONDARY OUTCOMES:
Stool frequency | 4 weeks
  Assessed by daily parental reporting.
Stool amount and stool colour | 4 weeks
  Assessed by the parents in a continuous daily bowel diary over the study period using the Amsterdam Infant Stool Scale (AISS). Stool amount will be assessed on a 4-point scale (1: smear, 2: up to 25%, 3: 25.50%, 4: >50%, relative to diaper surface). Stool colour will be assessed on a 6-point scale (I: yellow, II: orange, III: green, IV: brown, V: meconium, VI: clay-coloured)
Treatment success | 4 weeks
  ROME IV criteria still met at the end of the intervention.
Faecal microbiota | 4 weeks
  Stool samples will be analyzed by appropriate molecular biological methods like 16S rRNA gene sequencing to gain insight into the composition of the gut microbiota. Furthermore, metabolites like SCFA and other organic acids will be measured with appropriate chromatographic methods.
Faecal Short Chain Fatty Acids concentration | 4 weeks
  Change in Short Chain Fatty Acids over a four week period.
Faecal pH | 4 weeks
  Change in faecal pH over a four week period.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Cai, Doctor, Principal Investigator — Xin Hua Hospital，School of Medicine, Shanghai Jiaotong University; Weihui Yan, Doctor, Study Director — Xin Hua Hospital，School of Medicine, Shanghai Jiaotong University; Ying Wang, Doctor, Study Chair — Xin Hua Hospital，School of Medicine, Shanghai Jiaotong University; Lina Lu, Doctor, Study Chair — Xin Hua Hospital，School of Medicine, Shanghai Jiaotong University; YIjing Tao, Study Chair — Xin Hua Hospital，School of Medicine, Shanghai Jiaotong University; Haixia Feng, Study Chair — Xin Hua Hospital，School of Medicine, Shanghai Jiaotong University; Yinghong Chen, Study Chair — Xin Hua Hospital，School of Medicine, Shanghai Jiaotong University; Anna Li, Study Chair — Xin Hua Hospital，School of Medicine, Shanghai Jiaotong University
Locations (1):
- Shanghai Xinhua Hospital, affiliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Closa-Monasterolo R, Ferre N, Castillejo-DeVillasante G, Luque V, Gispert-Llaurado M, Zaragoza-Jordana M, Theis S, Escribano J. The use of inulin-type fructans improves stool consistency in constipated children. A randomised clinical trial: pilot study. Int J Food Sci Nutr. 2017 Aug;68(5):587-594. doi: 10.1080/09637486.2016.1263605. Epub 2016 Dec 8. PMID 27931142